CLINICAL TRIAL: NCT02718885
Title: Gut Microbiome Mediated Effects of Inulin Supplementation on Mineral and Bone Metabolism in Hemodialysis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Kenneth Wilund, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 16035
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Bone Diseases, Endocrine; Nutritional and Metabolic Diseases
Keywords: inulin-type fructans; hemodialysis; gut microbiome; mineral and bone disorder
MeSH Terms: conditions — Bone Diseases, Endocrine; Nutritional and Metabolic Diseases; Calcinosis; Bone Diseases | interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Sham Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin
- Inulin (Active Comparator): Inulin-type fructans
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Females will ingest 2 doses of 5g/inulin for a total of 10g/inulin/day for four weeks Males will ingest 2 doses of 7.5g/inulin for a total of 15g/inulin/day for four weeks
  Other Names: Inulin-type fructans
  Arms: Inulin
Dietary Supplement: Maltodextrin — Females will ingest 2 doses of 5g/maltodextrin for a total of 10g/maltodextrin/day for four weeks Males will ingest 2 doses of 7.5g/maltodextrin for a total of 15g/maltodextrin/day for four weeks
  Arms: Maltodextrin

SUMMARY:
The overall objective of the study is to examine the changes within the gut microbiome after the supplementation of inulin and its effect on markers of mineral metabolism and bone turnover.

DETAILED DESCRIPTION:
In this randomized controlled cross-over study, twenty HD patients (10 male/10 female, aged 20-80) will be recruited from local dialysis clinics in Champaign-Urbana, IL. After baseline testing, patients will be randomized to the intervention group or placebo group (maltodextrin). Patients will consume inulin (females 10g/day, males 15g/day) or maltodextrin (females 10g/day, males 15g/day) for one month, rest for two weeks (washout period), and continue with the other treatment (either inulin or maltodextrin) for another month. Outcomes will be assessed at the beginning of each period and after a month of supplementation at both periods.

ELIGIBILITY:
Inclusion Criteria:

* Receive HD therapy 3 days per week and for at least 3 months

Exclusion Criteria:

* Sustained hypercalcemia (>3months).
* Previous major gastrointestinal disease diagnosis (e.g., inflammatory bowel disease and celiac disease).
* Antibiotic treatment < 2 weeks prior the start of the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mineral metabolism | 4 weeks
  Plasma calcium, phosphorus and magnesium will be assessed by an blood-chemistry autoanalyzer at the beginning and end of each supplementation period. Additionally, parathyroid hormone and fibroblast-growth factor will be assessed by ELISA.

SECONDARY OUTCOMES:
Bone biomarkers | 4 weeks
  Sclerostin, bone-specific alkaline phosphatase and osteoprotegerin will be assessed by ELISA kits at the beginning and end of each period
Gut-microbiota derived metabolites | 4 weeks
  Free serum p-cresyl sulfate and indoxyl sulfate: serum (4ml) will be collected on midweek dialysis session and analyzed using an HPLC.
Gut microbiome | 4 weeks
  Participants will be asked to collect a complete fecal sample at the beginning and end of Period 1 and 2. V4 regions of the bacterial 16S rRNA gene will be isolated and amplified. Sequencing will be done through Illumina Mi-seq V3 platform. General changes in bacterial diversity and taxa will be analyzed through the open software QIIME.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wilund, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No